CLINICAL TRIAL: NCT07149402
Title: Serum Interleukin-33 (IL-33) Levels and Their Association With Clinical Manifestations in Patients With Systemic Lupus Erythematosus and Lupus Nephritis at Assiut University Hospital
Brief Title: Association of Serum Interleukin-33 Levels With Clinical Manifestations in Systemic Lupus Erythematosus
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marly Mamdouh, resident at the Rheumatology Department, Assiut University
Other Study IDs: SLE Interleukin-33 Levels
Record Dates: First submitted 2025-08-28; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: SLE
Keywords: SLE; IL-33

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLE without Nephritis: Patients diagnosed with systemic lupus erythematosus but without evidence of renal involvement. Clinical and laboratory data are collected to correlate IL-33 levels with disease activity excluding renal manifestations.
- SLE with Lupus Nephritis: Patients with systemic lupus erythematosus and confirmed lupus nephritis via biopsy and clinical parameters. This group undergoes detailed renal Doppler imaging and biopsy assessment to evaluate the relationship of IL-33 with renal involvement.
- Healthy Controls: Age- and sex-matched healthy individuals without autoimmune or renal disease, serving as baseline comparators for IL-33 serum levels and immune profiles.

SUMMARY:
This is a case-control study investigating serum IL-33 levels and their association with clinical manifestations in systemic lupus erythematosus (SLE). The study compares IL-33 levels in three groups: SLE patients with lupus nephritis, SLE patients without nephritis, and healthy controls. The goal is to clarify IL-33's role as a biomarker reflecting disease activity and organ involvement, especially renal pathology.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease with variable clinical presentations, ranging from mild symptoms to life-threatening organ damage. Lupus nephritis, a severe renal manifestation of SLE, significantly contributes to morbidity and mortality. IL-33, a cytokine from the IL-1 family, has been implicated in immune regulation and inflammation, emerging as a potential marker in SLE pathogenesis and progression.

This study systematically evaluates serum IL-33 levels in 96 participants divided into three groups: SLE patients with lupus nephritis, SLE patients without nephritis, and matched healthy controls. The study is conducted over one year at the Rheumatology Department of Assiut University Hospital. It includes clinical assessments, laboratory investigations (including ELISA for IL-33, autoantibody profiles, renal function), renal Doppler ultrasound for nephritis patients, and renal biopsy analyzed using ISN/RPS classification.

By assessing IL-33 levels alongside clinical manifestations, disease activity indices, and histopathological findings, the study aims to define IL-33's diagnostic and prognostic utility in lupus nephritis and overall SLE disease monitoring. Statistical analysis with SPSS includes ANOVA and correlation tests to detect differences and associations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Diagnosed with systemic lupus erythematosus according to the American College of Rheumatology (ACR) criteria.
* For the lupus nephritis group: confirmed diagnosis of lupus nephritis based on clinical, laboratory, and renal biopsy findings.
* For the control group: healthy individuals matched for age and sex, with no history of autoimmune or renal diseases.

Exclusion Criteria:

* Patients with other autoimmune diseases. Patients with chronic infections or malignancies. Pregnant or lactating women. Patients with end-stage renal disease (ESRD) or on dialysis. Individuals who refuse to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes three groups, each with 32 participants for a total of 96 individuals. Inclusion criteria for SLE patients consist of adults aged 18 to 65 years diagnosed per ACR criteria. The lupus nephritis group includes patients with biopsy-confirmed nephritis. Healthy controls are age- and sex-matched individuals without autoimmune or renal diseases.
  Exclusion criteria contain coexisting autoimmune diseases, chronic infections, malignancies, pregnancy or lactation, end-stage renal disease or dialysis, and those declining consent. This carefully selected population ensures reliable comparisons of IL-33 levels relative to clinical and pathological traits. The sample size was powered to detect medium effect size differences in IL-33 levels among the three groups.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-08-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum IL-33 levels | Baseline
  Quantification of serum IL-33 concentrations using a high-sensitivity ELISA kit across three groups: healthy controls, SLE patients without nephritis, and SLE patients with nephritis.

REFERENCES:
- [Background] Cayrol C, Girard JP. Interleukin-33 (IL-33): A nuclear cytokine from the IL-1 family. Immunol Rev. 2018 Jan;281(1):154-168. doi: 10.1111/imr.12619. PMID 29247993